CLINICAL TRIAL: NCT03450005
Title: ECMM Candida Registry - CandiReg
Acronym: CandiReg
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Prof. Dr. med., University of Cologne
Other Study IDs: Candi001
Record Dates: First submitted 2018-02-02; First posted 2018-03-01 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Invasive Candidiases
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fungal culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- emerging Candida isolates: Web-based registry of invasive infections by Candida species

SUMMARY:
The objective of the European Confederation of Medical Mycology - ECMM Candida Registry (CandiReg) is to overcome the lack of knowledge on epidemiology, clinical course, and molecular characteristics of invasive infections due to invasive Candida infections and to function as a platform for future studies and in case of outbreaks.

DETAILED DESCRIPTION:
The specific objectives are:

To describe the global incidence of invasive Candida infection To monitor trends globally and locally over time To define patient risk groups To assess antifungal resistance among Candida spp. causing invasive diseases worldwide To assess attributable mortality of invasive Candida infection To assess incremental costs associated with invasive Candida infection

To describe the clinical pattern of disease To document diagnostic procedures performed for confirmation of diagnosis To describe first-line and salvage treatment regimens applied, guideline adherence, their efficacy and impact on patient survival To inform consensus guidelines To develop clinical screening and diagnostic procedures

Set up of a collection of isolates with molecular characterization and evaluation of resistance genes

ELIGIBILITY:
Inclusion Criteria:

* Cultural, histopathological, antigen or DNA evidence of invasive fungal infection with Candida species.
* Hepatosplenic candidiasis with signs of disseminated Candida infection without culture, histological or microscopic evidence
* Case control

Matching procedure for controls:

In part, controls will be included at the same hospitals that include cases (i.e. each one control per case, both in the same hospital).

Controls will be matched by demographics, underlying diseases and risk factors as well as duration of hospitalization

Exclusion Criteria:

- Colonization or other non-invasive infection, including superficial skin infections, candiduria without dissemination or Candida spp. in stool.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasive infections caused by Candida species
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence | up to 100 weeks
  To describe the global incidence of invasive Candida infection
Mortality | up to 100 weeks
  To describe the global mortality of invasive Candida infection
Molecular characteristics of Candida auris | At 90 Days from diagnosis
  To describe the molecular characteristics of Candida auris
Susceptibility testing | At 90 Days from diagnosis
  To describe the susceptibility of Candida auris
Resistance development | up to 100 weeks
  To describe the resistance development of Candida auris

SECONDARY OUTCOMES:
Treatment efficacy of invasive candida infections | At 90 Days from diagnosis
  Number of participants with treatment failure
Treatment efficacy of invasive candida infections | At 90 Days from diagnosis
  Number of participants with stable disease
Treatment efficacy of invasive candida infections | At 90 Days from diagnosis
  Number of participants with partial response
Treatment efficacy of invasive candida infections | At 90 Days from diagnosis
  Number of participants with complete response

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, MD, Study Chair — University of Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany